CLINICAL TRIAL: NCT02261922
Title: A Prospective Randomized Double Blind Study to Evaluate the Effect of Ticagrelor on Endothelial Function
Brief Title: Ticagrelor and Endothelial Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hotel Dieu de France Hospital (Other)
Responsible Party: Principal Investigator, Rabih Azar, Chief of Cardiology, Hotel Dieu de France Hospital, Hotel Dieu de France Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FM240
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Antiplatelet Agents; Endothelial Function; Pleotropic Effects
MeSH Terms: interventions — Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ticagrelor (Experimental): ticagrelor treatment
  Interventions: Drug: ticagrelor
- prasugrel (Active Comparator): prasugrel treatment
  Interventions: Drug: prasugrel

INTERVENTIONS:
Drug: ticagrelor
  Arms: ticagrelor
Drug: prasugrel
  Arms: prasugrel

SUMMARY:
To evaluate the effect of ticagrelor on endothelial function as measured by flow mediated dilation of the brachial artery. This will be compared to prasugrel.

DETAILED DESCRIPTION:
Objective:

Demonstrate an improvement in endothelial function with ticagrelor

Introduction and hypothesis:

Ticagrelor and prasugrel are 2 new platelet antagonists. Both are superior to clopidogrel when used in acute coronary syndromes. However, only ticagrelor reduced cardiovascular mortality by almost 20%. Prasugrel reduced the composite clinical end point of cardiovascular mortality, myocardial infarction and stroke, but did not decrease mortality. The exact mechanism of mortality reduction with ticagrelor is unclear.

Some side effects of ticagrelor, such as brady-arrhythmias and dyspnea may be related to adenosine release. It is thus possible, that this drug may liberate significant amount of adenosine. Prior studies have demonstrated that adenosine has beneficial effects on the endothelial function and that it improves the outcome of patient with acute coronary syndromes.

It is thus possible that ticagrelor may improve endothelial function through an adenosine like effect. This effect is independent from platelet inhibition.

Prasugrel has the same platelet inhibition effect compared to ticagrelor, but our hypothesis is that it does not have an adenosine like effect and thus does not improve endothelial function.

Study design:

This is a prospective, randomized, double blind, cross-over study comparing 2 new platelet inhibitors that have the same potency: ticagrelor and prasugrel.

Patients with stable coronary artery disease will be randomized to one of these 2 drugs. Patients will receive one of the 2 drugs for a period of 8 +/- 2 days, they will then stop the drug for a period of 14 +/- 2 days, and they will then cross over and receive the other drug for a period of 8 +/- 2 days.

All patients will have the following measurements:

* Flow mediated Dilation (FMD) of the brachial artery
* Platelet aggregation in response to ADP

All measurements will be done at:

* Baseline 1 (prior to starting drug 1)
* At 8 +/- 2 days (peak effect of drug 1)
* Baseline 2 (at 14+/- 2 days; after washout and prior to starting drug 2)
* At 8 +/- 2 days after baseline 2 (peak effect of drug 2)

Measure of FMD of the brachial artery:

It will be performed according to the Academic Medical Center of Amsterdam pre-established protocol.

Measure of platelet aggregation:

It will be performed with the multiplate aggregometer

Study End-Points:

* Primary: change in FMD before and after each of the 2 drugs
* Secondary: Change in platelet aggregation before and after each of the 2 drugs
* Possible another secondary end-point: Change in NO activity in the blood before and after each of the 2 drugs

ELIGIBILITY:
Inclusion Criteria:

* - Prior MI > 1 year old
* Prior PCI > 1 year old
* Prior CABG > 3 months old
* Known lesion causing more than 50% stenosis on coronary angiography

Exclusion Criteria:

* Acute coronary syndrome within the last 6 months
* Any history of bleeding
* Age > 75 years
* Weight < 65 kg
* Prior stroke or TIA
* Platelet count < 100,000
* Hemoglobin < 11 mg/dL
* Patients who have received ticagrelor, prasugrel or clopidogrel in the 3 months that preceded randomization
* Patients who are taking anti-thrombotic therapy

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
flow mediated dilation of the brachial artery | 8 +/- 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hotel Dieu de France Hospital, El Achrafiyé, Beyrouth, Lebanon